CLINICAL TRIAL: NCT04287816
Title: Achieving Nutritional Adequacy Of Vitamin E With An Egg/Plant-Based Food Pairing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor and Principal Investigator, Ohio State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2019H0504-A
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Nutritional Requirements
Keywords: Vitamin E; Egg; Spinach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Zero hard-boiled egg at 0 h (Experimental): No eggs will be consumed on the test day. Deuterium-labeled spinach containing 5 mg αT will be ingested alone prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Zero hard-boiled egg at 0 h
- One hard-boiled egg at 0 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested along with 1 hard-boiled egg prior to the 72-h pharmacokinetics trial.
  Interventions: Other: One hard-boiled egg at 0 h
- Two hard-boiled eggs at 0 h (Experimental): Deuterium-labeled spinach containing 5mg αT will be ingested along with 2 hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Two hard-boiled eggs at 0 h
- Three hard-boiled eggs at 0 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested along with 3 hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Three hard-boiled eggs at 0 h
- One hard-boiled egg at 3 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested alone at 0 h prior to the 72-h pharmacokinetics trial followed by 1 hard-boiled egg 3 hours after spinach consumption.
  Interventions: Other: One hard-boiled egg at 3 h
- One hard-boiled egg at 0 h + One hard-boiled egg at 3 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested along with 1 hard-boiled egg at 0 h prior to the 72-h pharmacokinetics trial followed by 1 egg 3 hours after spinach consumption.
  Interventions: Other: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
- Two egg whites at 0 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested along with two egg whites prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Two egg whites at 0 h
- Vegetable oil at 0 h (Experimental): Deuterium-labeled spinach containing 5 mg αT will be ingested along with 9.6 grams of vegetable oil prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Vegetable oil at 0 h

INTERVENTIONS:
Other: Zero hard-boiled egg at 0 h — No eggs will be consumed on test day along with spinach consumption
  Arms: Zero hard-boiled egg at 0 h
Other: One hard-boiled egg at 0 h — One egg will be consumed on test day along with spinach consumption
  Arms: One hard-boiled egg at 0 h
Other: Two hard-boiled eggs at 0 h — Two eggs will be consumed on test day along with spinach consumption
  Arms: Two hard-boiled eggs at 0 h
Other: Three hard-boiled eggs at 0 h — Three eggs will be consumed on test day along with spinach consumption
  Arms: Three hard-boiled eggs at 0 h
Other: One hard-boiled egg at 3 h — One egg will be consumed on test day three hours after spinach consumption
  Arms: One hard-boiled egg at 3 h
Other: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h — Two eggs will be consumed on test day: one along with spinach consumption and the other one three hours after spinach consumption
  Arms: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
Other: Two egg whites at 0 h — Two egg whites will be consumed on test day along with spinach consumption
  Arms: Two egg whites at 0 h
Other: Vegetable oil at 0 h — 9.6 grams of Vegetable oil will be consumed on test day along with spinach consumption
  Arms: Vegetable oil at 0 h

SUMMARY:
Malnutrition of the fat-soluble nutrient vitamin E (α-tocopherol; αT) is problematic. Since αT is rich in plant foods (e.g. spinach) that are mostly absent of accessible lipid, dietary patterns that can potentiate αT bioavailability by pairing vegetables with lipid-rich foods have been emphasized. The purpose of this study is to use deuterium-labeled spinach (containing stable isotopes of αT) to validate eggs as a dietary tool to improve αT bioavailability directly from a model plant food, and hence achieve nutrient adequacy. It is expected that compared with deuterium-labeled spinach alone, co-ingestion of eggs will dose- and time-dependently increase plasma bioavailability of spinach-derived deuterium-labeled αT without affecting time to maximal concentrations or half-lives. Further, phospholipid-rich egg yolk lipid will enhance nutrient bioavailability compared with vegetable oil. The outcome will therefore support an egg-based food pairing that can enhance the health benefits of plant-centric dietary patterns.

DETAILED DESCRIPTION:
In the US, 92-96% of men and women do not meet recommended intakes for αT. Dietary recommendations strongly encourage a diet rich in fruits and vegetables to meet dietary αT requirements. However, αT bioavailability from most plant foods is quite poor, thereby emphasizing a need for effective food pairings that can enhance the absorption and promote adequate status of these health-promoting nutrients. The objective of this application is to use deuterium-labeled spinach (containing stable isotopes of αT) to validate eggs as a dietary tool to improve αT bioavailability directly from a model plant food, and hence achieve nutrient adequacy. Our hypothesis is that the bioavailability of αT from deuterium-labeled spinach will be potentiated by egg intake in a dose-dependent manner by increasing their secretion in intestinal-derived chylomicrons. Furthermore, phospholipid-rich whole eggs will enhance spinach-derived αT bioavailability compared with vegetable oil, and will be most functionally responsible for the benefits of eggs to enhance nutrient absorption. Additionally, egg whites will more greatly promote nutrient bioaccessibility compared with spinach alone.

To test this, our specific aim is to assess egg-mediated improvements in αT bioavailability by conducting a cross-over pharmacokinetic study in healthy men and women. In Study Arms 1-4, participants will ingest deuterium-labeled spinach (containing 5 mg αT) with 0, 1, 2, or 3 hardboiled eggs (containing 0, 4.8, 9.6, or 14.4 g total fat, respectively). In Study Arm 5, participants will ingest spinach with two egg whites. In Study Arm 6, participants will ingest spinach with 9.6 grams of vegetable oil. In Study Arm 5, participants will ingest spinach alone followed by 1 egg 3-hours later. In Study Arm 7, participants will ingest spinach with 1 egg followed by another egg 3-hours later. In Study Arm 8, participants will ingest spinach with 1 egg followed by another egg 3-hours later. Thus, Study Arms 1-6 will test the dose-dependent and food matrix effects of eggs on αT bioavailability, and study Arms 7-8 will test the meal timing effects of eggs on αT bioavailability. Eucaloric diets will be controlled for αT intakes for 3 d prior to and during the initial 24 h of each trial to minimize heterogeneity of pharmacokinetic responses. Spinach-derived deuterium-labeled αT will be measured in plasma and isolated chylomicrons collected at timed intervals from 0-72 h post-meal ingestion, and biomarkers of antioxidant status and oxidative distress will be assessed at baseline (0 h) of each trial. Outcomes from this study are expected to demonstrate a dose- and time-dependent function of eggs to increase deuterium-labeled αT bioavailability (based on area under the curve (AUC) 0-72 h, Cmax, and % estimated absorption).

The rationale for this study is that, by establishing the efficacy of eggs to potentiate plant-derived fat-soluble nutrient bioavailability, a strong framework will exist for an easily implementable health-promoting food pairing strategy to overcome malnutrition of αT.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) = 19-25 kg/m2
* Normolipidemic (total cholesterol <240 mg/dL; triglyceride <150 mg/dL)
* Fasting glucose <100 mg/dL
* Normal hematocrit level (41%-50% for men and 36%-48% for women)
* Normal hemoglobin level (13.5-17.5 g/dL for men and 12.0-15.5 g/dL for women)
* No use of dietary supplements for >1 month
* No use of medications that affect lipid or glucose metabolism
* Non-smoker
* No history of gastrointestinal disorders

Exclusion Criteria:

* Egg allergy
* Alcohol intake > 2 drinks per day
* Aerobic activity >7 h/wk
* Body mass change >2 kg in the past 1 month
* Women who are pregnant, lactating, or initiated or changed birth control in the past 3 month
* Vegetarian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bruno, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Participants received the following interventions in order across 8 periods:
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
- Sequence 2: Participants received one of the interventions listed in the periods. One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
- Sequence 3: Participants received one of the interventions listed in the periods. Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
- Sequence 4: Participants received one of the interventions listed in the periods. Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
- Sequence 5: Participants received one of the interventions listed in the periods. Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
- Sequence 6: Participants received one of the interventions listed in the periods. Vegetable oil at 0 h
  One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
- Sequence 7: Participants received one of the interventions listed in the periods. One hard-boiled egg at 3 h
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
- Sequence 8: Participants received one of the interventions listed in the periods. One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
  Zero hard-boiled egg at 0 h
  One hard-boiled egg at 0 h
  Two hard-boiled eggs at 0 h
  Three hard-boiled eggs at 0 h
  Two egg whites at 0 h
  Vegetable oil at 0 h
  One hard-boiled egg at 3 h
Period: SPINACH
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + 1 Egg (0 h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + 2 Eggs (0 h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + 3 Eggs (0 h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + WHITE
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + Oil
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Period: SPINACH + Egg (3 h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: SPINACH + Eggs (0 & 3 h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8
Started | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Completed | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics: Characteristics of participants upon enrollment into the study
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 21.8 (2.0)
Waist circumference Male [Mean (Standard Deviation); unit: cm] | 76.3 (4.2)
Waist circumference Female [Mean (Standard Deviation); unit: cm] | 74.1 (4.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 109.6 (8.3)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 70.8 (5.4)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.19 (0.47)
Triglyceride [Mean (Standard Deviation); unit: mmol/L] | 0.57 (0.15)
Total Lipid [Mean (Standard Deviation); unit: mmol/L] | 4.75 (0.57)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 4.81 (0.39)

OUTCOME MEASURES:

1. Primary Outcome: Vitamin E Area Under the Curve (0-72 h)
Description: Area under the concentration-time curve of plasma deuterium-labeled alpha-tocopherol over 72 hours post ingestion.
Time Frame: 0, 3, 4.5, 6, 7.5, 9, 12, 24, 36, 48, 72 hours post-ingestion of spinach
Measure: Mean (Standard Error); unit: umol/L*h
Groups:
- SPINACH: No eggs will be consumed on the test day. Deuterium-labeled spinach containing 5 mg alpha-tocopherol (αT) will be ingested alone prior to the 72-h pharmacokinetics trial.
  Zero hard-boiled egg at 0 h: No eggs will be consumed on test day along with spinach consumption
- SPINACH + 1 EGG0 h: Deuterium-labeled spinach containing 5 mg αT will be ingested along with 1 hard-boiled egg prior to the 72-h pharmacokinetics trial.
  One hard-boiled egg at 0 h: One egg will be consumed on test day along with spinach consumption
- SPINACH + 2 EGGS0h: Deuterium-labeled spinach containing 5mg αT will be ingested along with 2 hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Two hard-boiled eggs at 0 h: Two eggs will be consumed on test day along with spinach consumption
- SPINACH + 3 EGGS0 h: Deuterium-labeled spinach containing 5 mg αT will be ingested along with 3 hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Three hard-boiled eggs at 0 h: Three eggs will be consumed on test day along with spinach consumption
- SPINACH + WHITE: Deuterium-labeled spinach containing 5 mg αT will be ingested along with two egg whites prior to the 72-h pharmacokinetics trial.
  Two egg whites at 0 h: Two egg whites will be consumed on test day along with spinach consumption
- SPINACH + OIL: Deuterium-labeled spinach containing 5 mg αT will be ingested along with 9.6 grams of vegetable oil prior to the 72-h pharmacokinetics trial.
  Vegetable oil at 0 h: 9.6 grams of Vegetable oil will be consumed on test day along with spinach consumption
- SPINACH + EGG3 h: Deuterium-labeled spinach containing 5 mg αT will be ingested alone at 0 h prior to the 72-h pharmacokinetics trial followed by 1 hard-boiled egg 3 hours after spinach consumption.
  One hard-boiled egg at 3 h: One egg will be consumed on test day three hours after spinach consumption
- SPINACH + EGGS0 & 3 h: Deuterium-labeled spinach containing 5 mg αT will be ingested along with 1 hard-boiled egg at 0 h prior to the 72-h pharmacokinetics trial followed by 1 egg 3 hours after spinach consumption.
  One hard-boiled egg at 0 h + One hard-boiled egg at 3 h: Two eggs will be consumed on test day: one along with spinach consumption and the other one three hours after spinach consumption
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 5
umol/L*h | 2.90 (0.88) | 5.24 (1.00) | 5.18 (1.06) | 4.39 (0.69) | 5.10 (0.65) | 6.88 (0.74) | 1.67 (0.45) | 4.88 (1.53)

2. Primary Outcome: Vitamin E Cmax
Description: Maximum plasma concentration of deuterium-labeled alpha-tocopherol
Time Frame: 0-72 hours post-ingestion of spinach
Measure: Mean (Standard Error); unit: umol/L
Groups:
- SPINACH: No eggs will be consumed on the test day. Deuterium-labeled spinach containing 5 mg αT will be ingested alone prior to the 72-h pharmacokinetics trial.
  Zero hard-boiled egg at 0 h: No eggs will be consumed on test day along with spinach consumption
- SPINACH + 2 EGGS0 h: Deuterium-labeled spinach containing 5mg αT will be ingested along with 2 hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Two hard-boiled eggs at 0 h: Two eggs will be consumed on test day along with spinach consumption
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0 h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 5
umol/L | 0.09 (0.02) | 0.18 (0.03) | 0.15 (0.03) | 0.14 (0.02) | 0.15 (0.02) | 0.2 (0.02) | 0.06 (0.01) | 0.14 (0.04)

3. Secondary Outcome: Vitamin E Tmax (hr)
Description: Time to reach maximum plasma concentration of deuterium-labeled alpha-tocopherol
Time Frame: 0-72 hours post-ingestion of spinach
Measure: Mean (Standard Error); unit: hr
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0 h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 5
hr | 9.64 (0.86) | 10.10 (0.55) | 10.90 (0.55) | 9.94 (0.63) | 9.94 (0.63) | 9.38 (0.79) | 10.20 (0.74) | 9.90 (0.90)

4. Secondary Outcome: Half-Life (hr)
Description: The time required for the plasma concentration of vitamin E to decrease by 50%.
Time Frame: 0-72 hours post-ingestion of spinach
Measure: Mean (Standard Error); unit: hr
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 5
hr | 25.36 (4.54) | 22.52 (3.26) | 26.92 (2.25) | 24.34 (3.65) | 26.79 (1.57) | 30.45 (2.11) | 16.89 (2.53) | 21.24 (5.37)

5. Secondary Outcome: Estimated Absorption (%Dose) of Vitamin E
Description: Absorption of deuterium-labeled alpha-tocopherol
Time Frame: 0-72 hours post-ingestion of spinach
Measure: Mean (Standard Error); unit: Percent
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0 h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 5 | 5
Percent | 1.93 (0.50) | 3.52 (0.46) | 2.95 (0.53) | 2.96 (0.44) | 3.02 (0.44) | 3.86 (0.43) | 1.10 (0.22) | 2.70 (0.73)

6. Secondary Outcome: Chylomicron Vitamin E
Description: Deuterium-labeled alpha-tocopherol concentration in chylomicron
Time Frame: 0, 3, 4.5, 6, 7.5, 9, 12 hours post-ingestion of spinach
Population: Chylomicron measurements of vitamin E content were initially planned as part of the study protocol. While chylomicrons were isolated from blood samples and cryopreserved during the intervention, sample analysis was not performed because resources and personnel became unavailable. No data are available and these measures are not anticipated to be completed.
Arm/Group | SPINACH | SPINACH + 1 EGG0 h | SPINACH + 2 EGGS0 h | SPINACH + 3 EGGS0 h | SPINACH + WHITE | SPINACH + OIL | SPINACH + EGG3 h | SPINACH + EGGS0 & 3 h
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Primary Study: Participants (n = 8) completed six 72-hour pharmacokinetic trials in a crossover design. Each trial involved deuterium-labeled spinach (5 mg α-tocopherol) consumed at 0 h with one of the following:
  Spinach only (0 eggs)
  Spinach + 1 hard-boiled egg (0 h)
  Spinach + 2 hard-boiled eggs (0 h)
  Spinach + 3 hard-boiled eggs (0 h)
  Spinach + 2 egg whites (0 h)
  Spinach + vegetable oil (0 h) Trials were separated by ≥1-week washout. Spinach only (0 eggs, 0 h)
  Spinach + 1 hard-boiled egg (0 h)
  Spinach + 2 hard-boiled eggs (0 h)
  Spinach + 3 hard-boiled eggs (0 h) Spinach and 2 Eggs 0h Spinach and 3 Eggs 0h
- Exploratory Study: Participants (n = 5) completed two additional 72-hour pharmacokinetic trials in a crossover design, each separated by ≥1-week washout. Trials involved deuterium-labeled spinach (5 mg α-tocopherol) with:
  Spinach + 1 hard-boiled egg (3 h after spinach)
  Spinach + 1 hard-boiled egg at 0 h + 1 hard-boiled egg at 3 h.
  Spinach + 1 hard-boiled egg at 0 h + 1 hard-boiled egg at 3 h
  Spinach + 2 egg whites (0 h)
  Spinach + vegetable oil (0 h)
Arm/Group | Primary Study | Exploratory Study
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT04287816/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04287816/SAP_001.pdf
  • Informed Consent Form (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT04287816/ICF_002.pdf